CLINICAL TRIAL: NCT06715696
Title: Clinical Hemostatic Effectiveness of PET-Collagen Gauze ("HANBIO" Gauze) for Acute Wound: a Prospective, Single-arm, Open-label Evaluation Study
Brief Title: The Hemostatic Effectiveness of "HANBIO" Gauze During Non-emergent Gynecology Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAN Biomedical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HAN2018001-CT01
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Wounds and Injuries; Hemostasis
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- "HANBIO" Gauze (Experimental)
  Interventions: Device: "HANBIO" Gauze (Sterilized, 1% Collagen)

INTERVENTIONS:
Device: "HANBIO" Gauze (Sterilized, 1% Collagen) — After tissue resection in a standard procedure for gynecological surgery, direct application of "HANBIO" Gauze to cover the bleeding site/area which identified during dissection.

SUMMARY:
The objective of this study is to collect the hemostatic effectiveness and device safety data of "HANBIO" Gauze in subjects have acute wound result from gynecology surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female between 20 and 70 years of age.
* Subject scheduled for a non-emergent, gynecological surgery.
* Subject has an identified bleeding site/area intraoperatively.
* Subject is willing to comply with all aspects of the study and have signed informed consent form.

Exclusion Criteria:

* Pregnant or lactating female.
* The wound is chronic wound that not healed within 8 weeks, e.g. ulcers.
* The wound is caused by radiation or burns.
* Subject is sensitive or allergic to collagen.
* Subject is sensitive or allergic to polyester (PET).
* Subject has medical history of coagulation disorder or disease (e.g., hemophilia, thrombocytopenia).
* Subject receives anticoagulants or antiplatelets.
* Subject plans to receive other hemostatic gauze/dressing/agent/medical device as primary hemostasis.
* Subject has participated in another clinical trial within the past 30 days.
* Subjects with any pre-operative or intra-operative findings that may preclude conduct of the study procedure or unable to evaluate the outcomes.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Average Time(sec) to achieve hemostasis | 3 min
  The mean time(seconds) required to achieve hemostasis following the application of "HANBIO" Gauze.

SECONDARY OUTCOMES:
Proportions of subjects achieving hemostatic success at 3 min. | 3 min
  Subjects achieved success hemostasis within or at 3 minutes following the application of "HANBIO" Gauze.
Number/proportion of adverse and serious adverse events. | 3 min
  Subjects had AE or SAE following the application of "HANBIO" Gauze.
Ease of use questionnaire of Product "HANBIO" Gauze (by Principal Investigator) | 3 min
  Five questions regarding conveniency, non-adhesive property, conformability and hemostatic efficacy of "HANBIO" Gauze will be evaluated by surgeon(PI). One description, from "very satisfied", "satisfied", "neutral", "unsatisfied", "very unsatisfied", will be selected for each question.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan